CLINICAL TRIAL: NCT06064682
Title: An Organoid-based Functional Precision Medicine Trial in Osteosarcoma: PREMOST
Brief Title: An Organoid-based Functional Precision Medicine Trial in Osteosarcoma
Acronym: PREMOST
Status: Recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-001212
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-03

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: local tumor: patients with localized osteosarcoma who are scheduled to undergo diagnostic biopsy and are planned for surgical excision of the primary tumor
  Interventions: Other: standard of care biopsy
- Group 2: metastatic disease: patients with metastatic osteosarcoma who are scheduled to undergo either biopsy or surgery of metastatic disease
  Interventions: Other: standard of care biopsy

INTERVENTIONS:
Other: standard of care biopsy — Image-guided or surgical biopsy of the lesion that is suspected to be osteosarcoma in a patient with localized disease (Group 1)
  Groups: Group 1: local tumor
Other: standard of care biopsy — Image-guided or surgical biopsy or excision of the lesion that is suspected to be recurrent or metastatic osteosarcoma (Group 2).
  Groups: Group 2: metastatic disease

SUMMARY:
The purpose of this study is to examine if we can predict sensitivity of osteosarcoma to different chemotherapy agents using tissue cultures in the laboratory. We know that different chemotherapy agents can be used in the treatment, but not every sarcoma responds to them equally. It is important to understand if testing of the tissue obtained during a routine biopsy or surgery may be useful in selecting appropriate treatments. In addition, additional testing of the tumor, including genetic testing, will help us to understand osteosarcoma better.

DETAILED DESCRIPTION:
Investigators successfully established a miniaturized system that allows the setup of hundreds of wells and perform assays with minimal manipulation. The adapted geometry used to plate tumor cells in Matrigel, to generate mini-rings around the rim of the wells. This is attained by plating single-cell suspensions obtained from a cell line or a surgical specimen pre-mixed with cold Matrigel in a ring shape around the rim in 96-well plates. Rings can be established using a single-well or multichannel pipette. Cancer cell lines grown in mini-ring format give rise to organized tumor organoids that recapitulate features of the original histology. Treatment protocols and readouts for the mini-ring approach have been optimized. Seeding cells takes place on day 0, 2-3 days are allowed to establish organoids and it is followed by two consecutive daily drug treatments. The assay is flexible and can be easily adapted to single treatments followed by longer incubations, multiple consecutive recurring treatments, multi-drug combinations, or other screening strategies. Assays were implemented to quantify drug response by measuring cell viability after staining of live organoids with specific dyes followed by imaging. The pipeline has been extended to sarcomas: the team characterized organoids established from over 120 sarcoma biopsies, resections, and metastasectomies. Sarcoma organoids showed patient-specific growth characteristics and subtype-specific histopathology. Organoid sensitivity correlated with diagnostic subtype, patient age at diagnosis, lesion type, prior treatment history, and disease trajectory for a subset of the compounds screened. Organoid screening can provide information to facilitate optimal drug selection, avoid ineffective therapies, and mirror patient outcomes in sarcoma.

ELIGIBILITY:
Inclusion / exclusion criteria - Group1:

- Patients without diagnosis of osteosarcoma and whose imaging studies are suggestive of osteosarcoma and who are planned to undergo biopsy or surgery for diagnostic purposes

Inclusion / exclusion criteria - Group 2:

- Patients whose imaging studies are suggestive of metastatic osteosarcoma and who are planned to undergo biopsy or surgery for diagnostic purposes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Osteosarcoma is the most common primary bone malignancy of childhood and adolescence with a bimodal age distribution and a secondary peak in the 6th and 7th decades of life. The standard of care for localized disease is neoadjuvant cytotoxic chemotherapy followed by primary resection and adjuvant cytotoxic chemotherapy. Introduction of chemotherapy in the treatment of patients with osteosarcoma resulted in a significant improvement in the overall survival, but further improvement is needed.
  Currently, 5-year survival rate is 65 - 70%; for de novo metastatic disease or recurrent disease, 5-year survival rate is <30%. Recurrent or metastatic osteosarcomas are usually resistant to standard of care, and treatment options for refractory osteosarcomas are extremely limited.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
organoids from initial biopsy | two years
  To assess the feasibility of establishing organoids from initial biopsy and from postsurgical sample in patients with osteosarcoma, both in patients with localized disease and metastatic disease

SECONDARY OUTCOMES:
drug sensitivity of organoids | two years
  To compare drug sensitivity of organoids established from the original biopsy to drug sensitivity of organoids established from the surgical excision of the primary tumor after neoadjuvant chemotherapy
degree of necrosis in the tumor | two years
  To correlate the degree of necrosis in the tumor obtained by the surgical excision of the primary tumor after neoadjuvant chemotherapy with the chemotherapeutic drug sensitivity in the organoids.
clinical benefit | two years
  To correlate the magnitude of clinical benefit in patients with metastatic osteosarcoma treated with systemic chemotherapy with the chemotherapeutic drug sensitivity in the organoids established from biopsy or surgical excision of metastatic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Soragni, PhD, Principal Investigator — University of California at Los Angeles
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States